CLINICAL TRIAL: NCT04928768
Title: Factors Influencing Patient Satisfaction in an Egyptian Sample After Orthodontic Treatment of Different Malocclusions. An Observational Cross Sectional Study
Brief Title: Factors Influencing Patient Satisfaction in an Egyptian Sample After Orthodontic Treatment of Different Malocclusions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Abdallah Elfaisal AbdelHakam, Principal Investigator, Cairo University
Other Study IDs: 39012
Record Dates: First submitted 2021-06-07; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A validated questionnaire (five-point Likert scale) through 10 items developed by Lee et al 2018 is employed to measure the level of orthodontic treatment satisfaction in 10 items; overall satisfaction, tooth alignment, facial appearance, eating and chewing, confident smile and self-image, retention state, treatment duration, treatment costs, intention to recommend, and relief of previous concerns. Total satisfaction is calculated by averaging the Likert scores from the 10 items

SUMMARY:
Previously, patient satisfaction with orthodontic treatment has been reported at a broad range of 34% to 95% but these values mostly represent satisfaction for tooth alignment or simple satisfaction with treatment results. In keeping with the increased focus on patient satisfaction, many other factors were put into consideration in our study which contributes to the level of total satisfaction as host factors, concerns regarding the treatment, treatment motivation and discomfort during or after treatment. There are also a lack of studies conducted for orthodontic treatment satisfaction using previously validated questionnaires as well as correlation between patient's treatment satisfaction and ABO grading hasn't been sufficiently discussed in the literature, this study aims to address that gap. It would be also beneficial to investigate the frequency of different malocclusions presented in a sample of postorthodontic patients as it will give an insight about the distribution of the different malocclusion treated within the clinic and the degree of success in treating such malocclusions.

DETAILED DESCRIPTION:
Research Procedure in brief:

The following will be done for each participant:

Collection of patients telephone numbers:

Through the orthodontic department patient's database ensuring complete confidentiality. Telephoning the patients for follow ups after orthodontic treatment and asking them to fill in a questionnaire during their visit for explaining our aim for the study.

Personal data chart:

Including name, age, date of birth, mobile number and address. Examination of pretreatment records of the patients included in the sample to detect the type of malocclusion presented initially.

Orthodontic treatment satisfaction questionnaire:

The questionnaire is reviewed by faculty experts to determine whether the items in the questionnaire truly represent the items to be measured.

The translated questionnaire's face validation is led by the expert faculty members who are specialists in both English and Arabic guaranteeing clarity, intelligibility and comprehensiveness of items. This is significant in light of the fact that while performing any questionnaire in another setting, not all of the items may be compatible to Egyptian culture and lifestyles. In addition, a portion of items may not be applicable to specific age groups.

ABO Grading System Study models will be selected from the orthodontic department database. The post-treatment models will be assessed using the MGS of the American Board of Orthodontics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with different malocclusions who received and completed their fixed orthodontic treatment.
* Age: 16 years old or above.
* Patients who have completed their orthodontic treatment between November 2020 and November 2021.

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients below 16 years old.
* Illiterate patients.
* Patients who finished their treatment before November 2020 and after November 2021

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: male and female patients above 16 years with different malocclusion who recieved and completed their fixed orthodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall level of Orthodontic treatment satisfaction | 1 year
  unit of measurement: Likert Score form 1 to 5 (Qualitative- Ordinal)

SECONDARY OUTCOMES:
ABO grading of the finished cases | 1 year
  unit of measurement : ABO grading in points (Quantitative measures)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keles F, Bos A. Satisfaction with orthodontic treatment. Angle Orthod. 2013 May;83(3):507-11. doi: 10.2319/092112-754.1. Epub 2012 Nov 26. PMID 23181757
- [Background] Lee R, Hwang S, Lim H, Cha JY, Kim KH, Chung CJ. Treatment satisfaction and its influencing factors among adult orthodontic patients. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):808-817. doi: 10.1016/j.ajodo.2017.09.015. PMID 29853238
- [Background] Feldmann I, List T, John MT, Bondemark L. Reliability of a questionnaire assessing experiences of adolescents in orthodontic treatment. Angle Orthod. 2007 Mar;77(2):311-7. doi: 10.2319/0003-3219(2007)077[0311:ROAQAE]2.0.CO;2. PMID 17319767
- [Result] Al-Omiri MK, Abu Alhaija ES. Factors affecting patient satisfaction after orthodontic treatment. Angle Orthod. 2006 May;76(3):422-31. doi: 10.1043/0003-3219(2006)076[0422:FAPSAO]2.0.CO;2. PMID 16637722